CLINICAL TRIAL: NCT01953900
Title: Vaccination to Enhance the Anti-Tumor Activity of GD2 Chimeric Antigen Receptor-Expressing, VZV-Specific T Cells in Subjects With Advanced Sarcomas and Neuroblastoma (VEGAS)
Brief Title: iC9-GD2-CAR-VZV-CTLs/Refractory or Metastatic GD2-positive Sarcoma and Neuroblastoma
Acronym: VEGAS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Sarah Whittle, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-32335 VEGAS; VEGAS (Other: CAGT); P01CA094237 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Osteosarcoma; Neuroblastoma
Keywords: Osteosarcoma; T-Cells; varicella zoster virus (VZV); GD2; Neuroblastoma
MeSH Terms: conditions — Osteosarcoma; Neuroblastoma; Chickenpox | interventions — Herpes Zoster Vaccine; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GD2 T cells plus VZV vaccine (Experimental): In this study we will be administering from 1 x 10^6 to 1 x 10^9 transduced autologous VZV-specific CTLs, derived from VZV-specific memory T cells, so there will be no risk of alloreactivity. 6.1.1 Pre-infusion lymphodepletion for dose levels 9-11: Patients will receive 3 daily doses of cyclophosphamide together with fludarabine to induce lymphopenia, finishing at least 24 hours before T cell infusion. Cyclophosphamide will be given at a dose of 500 mg/m2/day followed by Fludarabine 30 mg/m2/day.
  Interventions: Genetic: GD2 T cells; Biological: VZV vaccine; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: GD2 T cells — On dose levels 1 and 2 each patient receives one injection of GD2 T cells followed by VZV vaccine injection 42 days later.
  Dose Level 1: 1x10^6 cells/m^2
  Dose Level 2: 1x10^7 cells/m^2
  The next dose levels to be studied following Dose level 2 are Dose levels 7 and 8 where subjects will receive the VZV vaccine followed by a single infusion of iC9-GD2-CAR-VZV-CTLs within 48 hours after VZV vaccine:
  Dose Level 7: 1 x 10^7 cells/m2
  Dose Level 8: 1 x 10^8 cells/m^2
  Dose levels 9-11 will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine prior to administration of the T cells.
  Dose Level 9: 1 x 10^8 cells/m^2
  Dose Level 10: 5 x 10^8 cells/m^2
  Dose Level 11: 1 x 10^9 cells/m^2
  The previously planned dose levels 3-6 will not be studied.
  Other Names: iC9-GD2-CAR-VZV-CTL
Biological: VZV vaccine — Subjects will receive a VZV vaccine with CTL infusion within 48 hours after the vaccine.
  Other Names: zostavax
Drug: Fludarabine — Pre-infusion lymphodepletion for dose levels 9-11: Patients will receive 3 daily doses of cyclophosphamide together with fludarabine to induce lymphopenia, finishing at least 24 hours before T cell infusion. Cyclophosphamide will be given at a dose of 500 mg/m^2/day followed by Fludarabine 30 mg/m^2/day. Infusions should be given following hospital/pharmacy recommendations however at a minimum the cyclophosphamide should be infused over 1 hour and the fludarabine should be infused over 30 minutes. Mesna, IV hydration, and anti-emetics will be provided following local institutional guidelines. T cell infusion will take place the day after completion of chemotherapy. Zostavax will be administered two weeks after infusion of T cells.
  Other Names: Fludara
Drug: Cyclophosphamide — Pre-infusion lymphodepletion for dose levels 9-11: Patients will receive 3 daily doses of cyclophosphamide together with fludarabine to induce lymphopenia, finishing at least 24 hours before T cell infusion. Cyclophosphamide will be given at a dose of 500 mg/m^2/day followed by Fludarabine 30 mg/m^2/day. Infusions should be given following hospital/pharmacy recommendations however at a minimum the cyclophosphamide should be infused over 1 hour and the fludarabine should be infused over 30 minutes. Mesna, IV hydration, and anti-emetics will be provided following local institutional guidelines. T cell infusion will take place the day after completion of chemotherapy. Zostavax will be administered two weeks after infusion of T cells.
  Other Names: Cytoxan

SUMMARY:
The purpose of this study is to find the largest safe dose of GD2-T cells (also called iC9-GD2-CAR-VZV-CTLs) in combination with a varicella zoster vaccine and lymohodepleting chemotherapy. Additionally, we will learn what the side effects of this treatment are and to see whether this therapy might help patients with advanced osteosarcoma and neuroblastoma. Because there is no standard treatment for recurrent/refractory osteosarcoma and neuroblastoma at this time or because the currently used treatments do not work fully in all cases, patients are being asked to volunteer to take part in a gene transfer research study using special immune cells.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise, but have not been strong enough to cure most patients.

Investigators have found from previous research that a new gene can be put into T cells that will make them recognize cancer cells and kill them. Investigators now want to see if a new gene can be put in these cells that will let the T cells recognize and kill sarcoma and neuroblastoma cells. The new gene is called a chimeric antigen receptor (CAR) and consists of an antibody called 14g2a that recognizes GD2, a protein that is found on sarcoma and neuroblastoma cells (GD2-CAR). In addition, it contains parts of the CD28 and OX40 genes which can stimulate T cells to make them live longer.

Investigators have found that CAR-T cells can kill some of the tumor, but they don't last very long in the body and so the tumor eventually comes back. T cells that recognize the virus that causes chicken pox, varicella zoster virus (VZV), remain in the bloodstream for many years especially if they are stimulated or boosted by the VZV vaccine. Investigators will therefore insert the GD2-CAR gene into T cells that recognize VZV. These cells are called iC9-GD2-CAR-VZV-specific T cells but are referred to as GD2-T cells for simplicity.

DETAILED DESCRIPTION:
Patients give blood to make GD2-T cells that are grown and frozen. To get the GD2-CAR to attach to the surface of the T-cell, a gene is inserted into the T-cell. As described in the Brief Summary, the gene contains the GD2-CAR. This is done using part of a virus (known as a retrovirus) that has been put into a vector made for this study and that will carry the antibody gene into the T cell. This retrovirus vector also helps identify the T cells in the patient's blood after they have been injected. Because the patients have received cells with a new gene in them they will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

When enrolled on this study, patients will be assigned to one of three groups of different doses of GD2-T cells. The first group of patients will receive a lower dose of GD2-T cells. Once that dose schedule proves safe, the next group of patients will be started at the higher dose. Patients will receive treatment with with cyclophosphamide (cytoxan) and fludarabine for 3 days before receiving the T-cell infusion. These drugs will decrease the numbers of your own T cells before we infuse the GD2-T cells.

Patients will receive the GD2-T cells by an intravenous line. Before patients receive the injection, they may be given a dose of Benadryl and Tylenol. The injection will take between 1 and 25 minutes. The research team will follow patients in the clinic after the injection for 1 to 4 hours. Two weeks after receiving the dose of GD2-T cells, patients will receive a dose of the VZV vaccine. This will be given as an injection under the skin that will take less than a minute. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital. Patients may need to stay in Houston for up to 4 weeks after the infusion so the research team can monitor patients for side effects. The research team will follow patients in the clinic or through communication with their primary doctor after the GD2-T-cell injection.

Medical tests before treatment--

Before being treated, patients will receive a series of standard medical tests:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function
* A urine pregnancy test. If you a patient is pregnant, both the patient and her parents will be informed of the pregnancy
* Measurements of their tumor by routine imaging studies. We will use the imaging study that was used before to follow the patient's tumor (Computer Tomogram (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography(PET/CT)

Medical tests during and after treatment--

Patients will receive standard medical tests when they are getting the infusions and afterwards:

* Physical exams
* Blood tests to measure blood cells, kidney and liver function
* Measurements of their tumor by routine imaging studies at 6 weeks after the infusion

To learn more about the way the GD2-T cells are working and how long they last in the body, an extra amount of blood, based on the patient's weight, up to a maximum of 60 ml (12 teaspoons) of blood will be taken on the day of the GD2-T- cell infusion(s), (before and at the end of the T-cell infusion(s)), 1, 2, 4, and 6 weeks after the GD2-T-cell infusion(s) and every 3 months for 1 year, at 15 months and 18 months, then every 6 months for 4 years, then yearly for a total of 15 years. One additional blood sample might be drawn 3 to 4 days after the GD2-T-cell infusion(s); this is optional. Blood may be drawn at additional time points based on the patient's response to the treatment.

During the time points listed above, if the Tcells are found in patient's blood at a certain amount, an extra 5ml of blood may need to be collected for additional testing.

For children, the total amount of blood drawn will not be more than 3 ml (less than 1 teaspoon) per 2.2 pounds of body weight on any one day. This volume is considered safe, but may be decreased if the patient is anemic (have a low red blood cell count).

ELIGIBILITY:
Inclusion Criteria:

Procurement:

* Diagnosis of relapsed or refractory osteosarcoma OR relapsed or refractory high risk neuroblastoma not responsive to standard treatment.
* Either previously infected with varicella zoster virus(VZV; chicken pox) or previously vaccinated with VZV vaccine
* Karnofsky/Lansky score of greater than or equal to 50
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Treatment:

* Diagnosis of relapsed or refractory osteosarcoma OR relapsed or refractory high risk neuroblastoma not responsive to standard treatment.
* Recovered from the acute toxic effects of all prior chemotherapy
* Karnofsky/Lansky score of greater than or equal to 50
* Bilirubin less than or equal to 3x upper limit of normal, AST less than or equal to 5x upper limit of normal, Serum creatinine less than or equal to 2x upper limit of normal, Hgb greater than or equal to 7.0 g/dl, ANC>500/uL, platelets > 50,000/uL
* Pulse oximetry of greater than or equal to 90% on room air
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the CTL infusion. Male partner should use a condom.
* Available autologous transduced cytotoxic T lymphocytes with greater than or equal to 20% expression of GD2 CAR and killing of GD2-positive targets greater than or equal to 20% in cytotoxicity assay
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria:

Procurement:

• Known primary immune deficiency or HIV positivity

Treatment:

* Severe intercurrent infection
* Known primary immune deficiency or HIV positivity
* Pregnant or lactating
* History of hypersensitivity reactions to murine protein-containing products
* Known allergy to VZV vaccine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2034-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity | 6-weeks
  The primary objective is to evaluate the safety and feasibility of intravenous injections of autologous iC9-GD2-CAR-VZV-CTLs in combination with VZV vaccination in patients with advanced GD2-positive sarcomas or neuroblastoma.

SECONDARY OUTCOMES:
Amount of T cells in the blood after the infusions | 15 years
  To assess the effects of VZV vaccination on the in vivo expansion and persistence of transgenic VZV-specific T cells
  To assess the in vivo persistence of infused T cells using immunoassays and transgene detection
Number of patients with a response to the T cells | 14 weeks
  To assess the anti-tumor effects of the infused GD2-specific T cells
  To assess the effect of of myeloid derived suppressor cells (MDSC) on expansion and persistence of infused T cells.
  Evaluations of tumor size will be performed within 4 weeks of beginning treatment and 6 weeks (before the vaccine) and 12 to 14 weeks after the iC9-GD2-CAR-VZV-CTL injection. All patients who receive the first infusion will be evaluable for response.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Wang, MD, Principal Investigator — Baylor College of Medicine; Sarah Whittle, MD, Principal Investigator — Pediatrics, Baylor College of Medicine; Cliona Rooney, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- [Derived] Tanaka M, Tashiro H, Omer B, Lapteva N, Ando J, Ngo M, Mehta B, Dotti G, Kinchington PR, Leen AM, Rossig C, Rooney CM. Vaccination Targeting Native Receptors to Enhance the Function and Proliferation of Chimeric Antigen Receptor (CAR)-Modified T Cells. Clin Cancer Res. 2017 Jul 15;23(14):3499-3509. doi: 10.1158/1078-0432.CCR-16-2138. Epub 2017 Feb 9. PMID 28183713